CLINICAL TRIAL: NCT06392269
Title: A Multi-site Clinical Evaluation of Capillary Blood Samples Collected Using the Tasso+SST Device for Downstream Analyte Testing.
Status: Recruiting | Type: Observational
Sponsor: Tasso Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: T23-02
Record Dates: First submitted 2024-04-07; First posted 2024-04-30 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Serum Analytes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum obtained from whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Tasso+: Comparison of capillary blood collected with a Tasso+ lancet vs. venous blood obtained via venipuncture
  Interventions: Diagnostic Test: Tasso+SST

INTERVENTIONS:
Diagnostic Test: Tasso+SST — Clinical evaluation of capillary blood samples collected using the Tasso+SST device for downstream analyte testing.

SUMMARY:
This is a prospective, multi-center study within the U.S. Study participants will take part in two study visits a minimum of 14 days apart. During each visit, participants will self-collect capillary blood samples. Additionally, a healthcare provide will obtain capillary and venous serum samples. All capillary samples will be collected from the upper arm using the Tasso+ device paired with a commercially-available serum separator gel microtainer. The samples will be shipped to a clinical laboratory and tested for various analytes. Expected analyte values for each participant will be based on their venous sample results which will be compared to Tasso sample results

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 - 85 years
2. Willing and able to provide written informed consent prior to study entry
3. Willing and able to adhere to study assessments, schedule, prohibitions and restrictions as described in the protocol
4. Healthy individuals or patients with analyte values (verified or likely to be) within intended clinical reference ranges as indicated by standard of care testing and/or past medical history (which may be documented or self-reported)

Exclusion Criteria:

1. Present with abnormal skin integrity or atypical skin health near/on arm collection sites
2. Mental or physical impairment which would preclude participation in the judgement of the investigator or qualified designee
3. Laboratory and healthcare personnel.
4. Any condition which, in the opinion of the Investigator or delegate, makes the participant unsuitable for this study (including, but not limited to, any mental or physical impairment which would preclude provision of adequate and knowledgeable consent)

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy individuals or patients with analyte values (verified or likely to be) within intended clinical reference ranges as indicated by standard of care testing and/or past medical history
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Number participants for which there is statistical concordance between serum biomarker results obtained from capillary blood vs. venous blood | 2 Weeks
  To establish the clinical performance of the Tasso+SST device for lay user self-collection and for trained healthcare provider (HCP) collection of capillary blood samples for downstream analyte testing at a clinical laboratory.

SECONDARY OUTCOMES:
Number of lay users in a simulated home setting for with statistical concordance between serum biomarker results obtained from capillary blood vs. venous blood | 1 Day
  To evaluate the performance of Tasso+SST capillary samples collected by lay users in a simulated home environment
Number of observed device usability issues observed in lay users and HCP populations, i.e., deviations from the instructions for use. | 2 Weeks
  To demonstrate usability of the Tasso+SST device in naive lay users and in trained HCP populations
Number participants for which there is statistical concordance between serum biomarker results obtained from Tasso+ capillary blood by two different HCPs | 2 weeks
  To demonstrate HCP inter-operator precision of Tasso+SST samples
Number participants for which there is statistical concordance between serum biomarker results obtained from Tasso+ capillary blood by the same lay user | 2 Weeks
  To demonstrate lay user intra-operator precision of Tasso+SST samples

CONTACTS AND LOCATIONS:
Locations (1):
- Tasso Research Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Research results are proprietary; no sharing with other researchers is anticipated.